CLINICAL TRIAL: NCT01942174
Title: Lead Time of the Methotrexate Establishment and Vaccinal Protection Against the Pneumococcal Agent in Patients Affected With Rheumatoid Polyarthritis
Brief Title: VACcination In Methotrexate Treated Rheumatoid Arthritis Patients
Acronym: VACIMRA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Hôpital Cochin (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9144
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Antipneumococcal vaccination; Methotrexate treatment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — 13-valent pneumococcal vaccine; Pneumococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate group (Other): For these patients, the methotrexate treatment is initiated in the same time that the antipneumococcal vaccination by Prevenar13. A revaccination by Pneumo23/Pneumovax is administred 2 months after the first vaccination.
  Interventions : biological/vaccine and drug
  Interventions: Biological: Prevenar 13; Biological: Pneumo23 / Pneumovax; Drug: Methotrexate - Immediate
- period group (Experimental): Methotrexate treatment is initiated 1 month later the first antipneumococcal vaccination by Prevenar13.
  A revaccination by Pneumo23/Pneumovax is administred 2 months after the first vaccination
  Interventions : biological/vaccine and drug
  Interventions: Biological: Prevenar 13; Biological: Pneumo23 / Pneumovax; Drug: Methotrexate - Delay

INTERVENTIONS:
Biological: Prevenar 13 — Vaccination at the beginning of the study (day 0)
  Other Names: Antipneumococcal vaccination
Biological: Pneumo23 / Pneumovax — Vaccination 2 months later the beginning of the study NB : Vaccine Pneumo23 has been replaced by equivalent vaccine Pneumovax in September 2017 because of the stop of commercialization of Pneumo23 in France by the pharmaceutical company
  Other Names: Antipneumococcal vaccination
Drug: Methotrexate - Immediate — concerning immediate group, methotrexate is Initiated in the same time that the antipneumococcal vaccination by prevenar 13
  Other Names: conventional methotrexate treatment
  Arms: Immediate group
Drug: Methotrexate - Delay — For "period group", methotrexate is Initiated & month after the antipneumococcal vaccination by prevenar 13
  Other Names: Experimental methotrexate treatment
  Arms: period group

SUMMARY:
To estimate the rate of immunological answer 1 month after antipneumococcal vaccination by the conjugated vaccine Prevenar13 ® in patients suffered from rheumatoid polyarthritis and who begin a treatement by methotrexate either in the same time, either 1 month later.

DETAILED DESCRIPTION:
Patients suffering from rheumatoid polyarthritis have an increased risk to develop an infection compared to general population, with a more important mortality risk because pneumococcus is considered as one of the major pathogenic agents. Antipneumcoccal vaccination is recommended to patients suffering from chronic inflammatory rheumatism treated with immunosuppressants. Methotrexate is a long term treatment used in first intention for rheumatoid polyarthritis. A recent study shows a decrease of efficacity of antipneumoccal vaccination for patients suffering from rheumatoid polyarthritis treated by methotrexate. The tested hypothesis will be the presence of better vaccinal protection for patients suffered from rheumatoid polyarthritis after 1 month between antipneumococcal vaccination and the initiation of methotrexate. The objective is to compare immunologic response for antipneumococcal vaccination between patients who are vaccinated in the same time of initiation of methotrexate and patients who are vaccinated 1 month before the beginning of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yeas old) suffers from rheumatoid arthritis considering ACR/EULAR 2010 criteria
* Rheumatoid arthritis considering 3,2<DAS<5,1
* Patient did not treat by long term treatment or has stopped a treatment by sulfasalazine, hydroxychloroquine or methotrexate for at least 3 months
* Patient has never treated by biotherapy
* Patient has never vaccinated against pneumococcal
* Patient has signed study consent form

Exclusion Criteria:

* Patient has ever treated by leflunomide or has treated previously by leflunomide (last 3 months)
* Patient is currently treated by methotrexate or has treated previously by methotrexate (last 3 months)
* Contraindication to methotrexate: renal insuffisance, alcoolic, chronic hepatisis, infectious condition, AIDS, hematological failure (cytopeny), pregnancy, obesity, diabet, respiratory disease, gastric ulcer
* Contraindication to corticotherapy
* Pregnancy or pregancy wish
* Nursing
* Absence of oral contraception for women of childbearing age
* Patient of age protected by law et deprived of liberty
* Subject who refuses to be vaccinated against pneumococcis agent
* Previous history of vaccination allergy (anaphylactic shok, Quincke oedema...)
* Gluten hypersensivity or intolerance
* Other vaccination during the last month before inclusion
* Ig perfusion during the last 3 months period before the study inclusion or during the study duration
* Patient currently treated by anticoagulant or has not been stopped for at least 48h before the study inclusion or hemostasis failure which is contraindicated with muscular injection
* Participation with an other clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
rate of immunological positive answer 1 month after antipneumococcal vaccination by the conjugated vaccine Prevenar13 ® in patients suffering from rheumatoid polyarthritis. | 1 month
  Patient who begins a treatement by methotrexate either in the same time, either 1 month later.
  An answer will be considered as positive if the patient answers in at least 3 on 5 of interest serotypes.

SECONDARY OUTCOMES:
Number of patients in each group who will know fully immunological answer to 5 interest serotypes after the first antipneumococcal vaccination (Prevenar13) | 1 month
Number of patients in each group who will know an immunological answer to 13 serotypes after the first antipneumococcal vaccination (Prevenar13) | 1 month
Number of patients who will know a fully immunological answer (13 serotypes of vaccine) after a antipneumococcal revaccination with Pneumo 23. | 3, 6 and 12 months
Number of patients who will suffer from adverse events in relation with the antipneumococcal vaccination | up to 12 months
Frequency of occurence of disease spurts from the first vaccination until the end of the study | Up to 12 months
occurence of the pneumococcal disease from the first vaccination to the end of the study. | 1, 6, 7 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacques MOREL, PU-PH, Principal Investigator — University Hospital, Montpellier
Locations (21):
- France (20):
  - CHU Nord, Amiens
  - CHU Pellegrin, Bordeaux
  - CHU La Cavale Blanche, Brest
  - CHU Montpied, Clermont-Ferrand
  - CHU Bicetre, Le Kremlin-Bicêtre
  - CH Du Mans, Le Mans
  - CHU Dupuytren, Limoges
  - CHU La Conception, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nice - Hôpital L'Archet 1, Nice
  - CHU Carémeau, Nîmes
  - CHU Orléans - Hôpital La Source, Orléans
  - CHU Saint Antoine, Paris
  - CHU La Pitié Salpétrière, Paris
  - CHU de Rennes, Rennes
  - CHU Bois Guillaume, Rouen
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - CHU Hautepierre, Strasbourg
  - CHU Purpan, Toulouse
  - CHU Trousseau, Tours
- CHPG Monaco - Hôpital Prince Grace de Monaco, Monaco, Monaco

REFERENCES:
- [Derived] Morel J, Dernis E, Roux C, Richez C, Brocq O, Fautrel B, Salliot C, Vittecoq O, Mariette X, Liote F, Lassoued S, Gaujoux-Viala C, Constantin A, Soubrier M, Devauchelle-Pensec V, Goeb V, Gottenberg JE, Marotte H, Moulard AR, Daien C, Mouterde G, Lukas C, Pissarra J, Huguet H, Launay O, Galtier F, Picot MC; I-REIVAC; CRI-IMIDIATE French Clinical Research Networks. Effect of a 1-month methotrexate delay on pneumococcal vaccine immunogenicity and disease control in patients with early rheumatoid arthritis (VACIMRA): an open-label randomised trial. Lancet Rheumatol. 2025 Oct;7(10):e675-e686. doi: 10.1016/S2665-9913(25)00071-2. Epub 2025 Jul 29. PMID 40749694